CLINICAL TRIAL: NCT03337191
Title: Ultrasound-Guided Versus Conventional Injection for Caudal Block in Children
Brief Title: Ultrasound-Guided Versus Conventional Injection for Caudal Block
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ataturk University (Other)
Responsible Party: Principal Investigator, Ali Ahiskalioglu, Principal Investigator, Ataturk University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: Caudal Ataturk Uni
Record Dates: First submitted 2017-11-06; First posted 2017-11-08 (Actual); Last update posted 2017-11-09 (Actual); Status verified 2017-11

CONDITIONS: Ultrasound Therapy; Complications
Keywords: ultrasound guided caudal injection; sacral hiatus; sacral canal
MeSH Terms: interventions — Levobupivacaine; Morphine; Ultrasonography

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- ultrasound guided caudal block (Active Comparator): Caudal block was performed by ultrasound guided with %0,125 levobupivacaine + 10 mq/kg morphine
  Interventions: Drug: Levobupivacaine; Drug: Morphine Sulfate; Device: Ultrasound
- conventional caudal block (Active Comparator): Caudal block was performed by conventional method with %0,125 levobupivacaine + 10 mq/kg morphine
  Interventions: Drug: Levobupivacaine; Drug: Morphine Sulfate

INTERVENTIONS:
Drug: Levobupivacaine — % 0,125 levobupivacaine
  Other Names: ultrasound guided caudal block
Drug: Morphine Sulfate — 10 mq/kg morphine sulfate
Device: Ultrasound — Ultrasound guided caudal block
  Arms: ultrasound guided caudal block

SUMMARY:
Caudal epidural block has been widely used, especially in pediatric surgery, to provide intraoperative and postoperative analgesia by affecting the region between T10 and S5 dermatomes in surgeries below the umbilical level.

In conventional single-shot caudal block, the needle is inserted through the skin with a 60-80 degrees angle, until the sacrococcygeal ligament is passed through. Then the angle of the needle is decreased to 20-30 degrees and inserted further for an additional 2-3 mm, entering into the sacral canal.There is a risk of dural or vascular puncture when the needle is passing through sacral canal. Other complications are the soft tissue bulging, intraosseous injections and systemic toxicity.

Many anatomical variations have been reported for sacral hiatus and sacral cornua. Therefore, the success rate of the classic caudal epidural anesthesia method in pediatric patients has been reported to be about 75%.

With the usage of ultrasonography in regional anesthesia, many advantages have been reported. Ultrasonography is helpful for visualization of the sacral hiatus, sacrococcygeal ligament, duramater, epidural space and the distribution of the local anesthetic agent within the epidural space. Therefore, this significantly increases the block success.

The primary aim of this study was compare the success rate of ultrasound guided sacral hiatus injection and conventional sacral canal injection. Secondary objectives are; block performing time, number of needle puncture, success at first puncture and complication rate.

ELIGIBILITY:
Inclusion Criteria:

* American Society of Anesthesiologist's physiologic state I-II patients undergoing phimosis and circumcision surgery

Exclusion Criteria:

* children with severe systemic disease
* previous neurological or spinal disorder,
* coagulation anomaly
* allergy against local anesthetics
* local infection at block site or
* with a history of premature birth

Ages: 5 Years to 12 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Child
Enrollment: 134 (Actual)
Dates: Start 2016-01-01 (Actual); Primary Completion 2016-07-01 (Actual); Study Completion 2016-09-01 (Actual)

PRIMARY OUTCOMES:
success rate of block | Intraoperative first hour
  A successful block was defined as absence of significant motor movements following surgical induction or heart and respiratory rates increasing not more than 20% of the basal levels.

SECONDARY OUTCOMES:
block performing time | Intraoperative first hour
  The block time was defined as the period between the insertion of the needle and termination of local anesthetic administration
first puncture success rate | Intraoperative first hour
  The first puncture success rate was defined as reaching the sacral canal or sacral hiatus with a single-needle orientation on the first puncture without any withdrawal from the skin.

CONTACTS AND LOCATIONS:
Locations (1):
- Ataturk University, Erzurum, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Dostbil A, Gursac Celik M, Aksoy M, Ahiskalioglu A, Celik EC, Alici HA, Ozbey I. The effects of different doses of caudal morphine with levobupivacaine on postoperative vomiting and quality of analgesia after circumcision. Anaesth Intensive Care. 2014 Mar;42(2):234-8. doi: 10.1177/0310057X1404200211. PMID 24580390
- [Background] Wang LZ, Hu XX, Zhang YF, Chang XY. A randomized comparison of caudal block by sacral hiatus injection under ultrasound guidance with traditional sacral canal injection in children. Paediatr Anaesth. 2013 May;23(5):395-400. doi: 10.1111/pan.12104. Epub 2012 Dec 29. PMID 23278906